CLINICAL TRIAL: NCT04842682
Title: A Phase I Multicenter Double-blind Placebo Controlled Dose Escalation Trial of an Adjuvanted Anti-CD40 mAb Fused to Env GP140 HIV Clade C ZM-96 (CD40.HIVRI.Env) Vaccine Combined or Not With a DNA-HIV-PT123 HIV-1 Vaccine in Healthy Participants
Brief Title: Dose Escalation Trial of CD40.HIVRI.Env Vaccine Combined or Not With a DNA-HIV-PT123 HIV-1 Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-001814-40; ANRS VRI06 (Other: ANRS)
Record Dates: First submitted 2021-03-24; First posted 2021-04-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Multicenter double-blind placebo controlled phase I dose-escalation trial to evaluate different dose levels of CD40.HIVRI.Env (adjuvanted with Hiltonol®) alone and in co-administration with DNA-HIV-PT123
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Within each group, participants will be randomized in a double blind manner to active intervention or placebo in a 5:1 ratio. Randomization will be stratified by group.
  All groups will be double-blind until W6. Formal individual unblinding (with communication of individual volunteer allocation to active vs. placebo) will only performed at the end of the W48 visits of all participants in a given group.
  Long term follow-up to study the persistence of immune responses at W76 will be unblinded.
  The second part of the trial will be single blind. Allocation of the use of the unadjuvanted vs. adjuvanted CD40. HIVRI.Env boost will be randomized. Randomisation will be stratified by the initial group (Solo or Combi with its dose level).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Active intervention (Experimental): Solo groups : CD40.HIVRI.Env vaccine (solution at 5.0 mg/ml) adjuvanted with Poly-ICLC (Hiltonol, solution at 1.8 mg/ml)
  Combi groups : CD40.HIVRI.Env vaccine (solution at 5.0 mg/ml) adjuvanted with Poly-ICLC (Hiltonol, solution at 1.8 mg/ml) and combined with DNA-HIV-PT123 HIV-1 vaccine (solution at 4.0 mg/ml)
  Interventions: Biological: Solo 0.3 group; Biological: Solo 1 group; Biological: Solo 3 group; Biological: Combi 0.3 group; Biological: Combi 1 group; Biological: Combi 3 group
- Part 1: Placebo (Placebo Comparator): Commercial Sodium Chloride at 0.9% (NaCl 0.9%)
  Interventions: Biological: Solo 0.3 group; Biological: Solo 1 group; Biological: Solo 3 group; Biological: Combi 0.3 group; Biological: Combi 1 group; Biological: Combi 3 group
- Part 2: Active intervention (Experimental): CD40.HIVRI.Env vaccine (solution at 5.0 mg/ml) adjuvanted or not with Poly-ICLC (Hiltonol, solution at 1.8 mg/ml)
  Interventions: Biological: Late boost CD40 alone; Biological: Late boost CD40 adjuvanted

INTERVENTIONS:
Biological: Solo 0.3 group — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 0.3 and 1.0 mg/injection, i.e. 1 ml subcutaneous route in right deltoid at weeks 0, 4 and 24
  Or, NaCl at 0.9%, i.e 1 ml subcutaneous route in right deltoid at weeks 0, 4 and 24.
  Arms: Part 1: Active intervention; Part 1: Placebo
Biological: Solo 1 group — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 1.0 and 1.0 mg/injection, i.e. 1 ml subcutaneous route in right deltoid at weeks 0, 4 and 24
  Or, NaCl at 0.9%, i.e 1 ml subcutaneous route in right deltoid at weeks 0, 4 and 24.
  Arms: Part 1: Active intervention; Part 1: Placebo
Biological: Solo 3 group — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 3.0 and 1.0 mg/injection, i.e. 1.2 ml subcutaneous route in right deltoid at weeks 0, 4 and 24
  Or, NaCl at 0.9%, i.e 1.2 ml subcutaneous route in right deltoid at weeks 0, 4 and 24.
  Arms: Part 1: Active intervention; Part 1: Placebo
Biological: Combi 0.3 group — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 0.3 and 1.0 mg/injection, i.e. 1 ml subcutaneous route in right deltoid; and combined with DNA-HIV-PT123 HIV-1 at 4.0 mg/injection, i.e. 1 ml intramuscular route in left deltoid at weeks 0, 4 and 24
  Or, NaCl at 0.9%, i.e 1 ml subcutaneous route in right deltoid and 1 ml intramuscular route in left deltoid at weeks 0, 4 and 24.
  Arms: Part 1: Active intervention; Part 1: Placebo
Biological: Combi 1 group — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 1.0 and 1.0 mg/injection, i.e. 1 ml subcutaneous route in right deltoid; and combined with DNA at 4.0 mg/injection, i.e. 1 ml intramuscular route in left deltoid at weeks 0, 4 and 24
  Or, NaCl at 0.9%, i.e 1 ml subcutaneous route in right deltoid and 1 ml intramuscular route in left deltoid at weeks 0, 4 and 24.
  Arms: Part 1: Active intervention; Part 1: Placebo
Biological: Combi 3 group — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 3.0 and 1.0 mg/injection, i.e. 1.2 ml subcutaneous route in right deltoid; and combined with DNA at 4.0 mg/injection, i.e. 1 ml intramuscular route in left deltoid at weeks 0, 4 and 24
  Or, NaCl at 0.9%, i.e 1.2 ml subcutaneous route in right deltoid and 1 ml intramuscular route in left deltoid at weeks 0, 4 and 24.
  Arms: Part 1: Active intervention; Part 1: Placebo
Biological: Late boost CD40 alone — CD40.HIVRI.Env at 0.3 mg/injection, i.e. 1 ml subcutaneous route in right deltoid at week LB (late boost)
  Arms: Part 2: Active intervention
Biological: Late boost CD40 adjuvanted — CD40.HIVRI.Env and Poly-ICLC (Hiltonol), respectively at 0.3 and 1.0 mg/injection, i.e. 1 ml subcutaneous route in right deltoid at week LB (late boost)
  Arms: Part 2: Active intervention

SUMMARY:
FIRST PART: DOSE ESCALATION Multicenter double-blind placebo controlled phase I dose-escalation trial that will be conducted in France and Switzerland to evaluate different dose levels of CD40.HIVRI.Env (adjuvanted with Hiltonol) alone and in co-administration with DNA-HIV-PT123.

A total of 72 eligible healthy participants will be recruited into 6 groups. Within each group, participants will be randomized in a double blind manner to active intervention or placebo in a 5:1 ratio. Enrolment into a given group (other than group "Solo 0.3") will open sequentially depending on the " go-criterion " based on the safety data of the preceding group(s).

The primary objective is to assess the safety of three dose levels of CD40.HIVRI.Env (0.3; 1; 3 mg) adjuvanted with Poly-ICLC (Hiltonol®), alone and in combination with DNA-HIV-PT123, administered at weeks 0, 4 and 24 in healthy participants.

Secondary objectives are to assess the capacity of poly-ICLC-adjuvanted CD40.HIVRI.Env alone and in combination with DNA-HIV-PT123 to elicit immune responses against HIV (immunogenicity):

* Humoral (antibody) responses ;
* B-cell responses ;
* T-cell responses.

SECOND PART: BOOST VACCINATION AND FOLLOW-UP Preliminary safety results allow consideration of long-term follow-up and evaluation of an additional CD40.HIVRI.Env booster injection in volunteers. An admendment was approved to complete the follow-up with two visits: 2 weeks (WLB+02) and 24 weeks (WLB+24) after the boost (WLB). Volunteers who received the active strategy in the first part of the trial (n=60) will be randomized in a single blind design and will receive an additional 0.3 mg dose of CD40HIVRI.Env vaccine either combined with Hiltonol adjuvant, as in the first part of the trial, or unadjuvanted. Part 2 will take place after the W48 visit and the participant's unblinding of Part 1.

It will address the following secondary objectives:

* To evaluate tolerance
* To evaluate the evolution of long-term vaccine responses (immunogenicity) and the effect of a booster injection of CD40.HIVRI.Env alone or adjuvanted with Poly ICLC- Hiltonol®. The tests that will be performed will be identical to those performed during the first phase of the trial allowing the monitoring of the evolution of responses.

DETAILED DESCRIPTION:
The ANRS VRI06 clinical trial follows the prophylactic vaccine strategies developed since the encouraging results obtained during the RV144 trial. The RV144 study identified binding IgG antibodies directed at conserved regions of the V1/V2 loop and antibody-dependent cell-mediated cytotoxicity as immune correlates of reduced risk of HIV infection in the absence of inhibiting serum IgA antibodies.

We have developed DC-targeting vaccines, in order to increase protein antigen efficacy through their selective delivery to dendritic cell (DC), the key cell type for initiating and regulating immune responses, via the endocytic receptors expressed at the DC surfaces. Following the screening of vaccines targeting different several DC-receptors, the CD40-targeting vaccine has been shown to be the best candidate for inducing both cellular and humoral responses. Anti-CD40.Env GP140 vaccine (CD40.HIVRI.Env) adjuvanted with Poly-ICLC (Hiltonol®), in a prime/boost association with poxvirus vector vaccines, has shown to be safe and elicit robust Env specific T and B cell responses in a non-human primate study.

In this trial we will also capitalize on data generated in a recent phase I/II trial showing that co-administration of DNA-HIV-PT123 with an Env protein vaccine (as compared to other vaccine regimens which do not co-administer the protein during the priming) results in the rapid generation of high titers of binding anti V1/V2 Env region IgG Abs and Tier 1 nAb responses (HVTN 096 study).

We therefore hypothesize that co-administration of CD40.HIVRI.Env adjuvanted with Poly-ICLC (Hiltonol®) with the DNA-HIV-PT123 vaccine will be safe and induce high titers of binding anti V1/V2 Env region IgG Abs and other immunological parameters considered as immune correlates in RV144 trial.

When the first 6 participants of given dose group have reached W6 (2 weeks after the second injection), the Protocol Safety Review Team (PSRT), composed of sponsor's pharmacovigilance expert, coordinating investigator, co-coordinating investigator and methodologist, will review all accumulated Adverse Event (AE) data so far, in a blinded manner. All AE, in particular grade 3 and grade 4 AEs, as well as Serious Adverse Events (SAEs) will be reviewed. The current version FDA grading scale will be used for grading.

Go-criterion for opening enrolment into the next groups: If no grade 3 or 4 clinical solicited local/systemic or unsolicited AE or grade 3 or 4 biological clinical significant, is reported at W6, in any of the first 6 participants of a given group, the Data and Safety Monitoring Board (DSMB) assessment will not be requested for the go to the next group and the " go-criterion " is met. The trial can be continued by opening to the inclusions following the protocol.

Otherwise (occurrence of grade 3 or 4 AE), the DSMB will review all accumulated AE data. Enrolment in next group will only start after the DSMB gives the green light.

In addition, the following pausing rule (pausing of all injections) will apply during the trial:

Pausing rule for vaccine related safety events : If a serious adverse reaction (relatedness as judged by the pharmacovigilance department or the investigator responsible of the SAE notification) is reported during any stage of the study, all vaccinations will be halted, inclusions in the trial will be suspended, competent authorities must be informed and an ad-hoc DSMB meeting convened for recommendations on the trial continuation. Vaccinations may resume only after authorization is given by competent authority.

By the conservative method, if the causality assessment could not be provided by the investigator, the AE will be considered as possibly related.

Based on the first safety and immunogenicity results, the study design has been amended with the addition of boost injection. Heterologous prime boost vaccination strategies in HIV have been associated with short-lived responses, notably in the RV144 trial, leading to the proposal of additional early boosts as in the RV702 trial or late boosts as in the RV305 trial. In the latter trial it was shown that only the boost with the protein component of the strategy was relevant in terms of restimulation of the immune response. Data obtained during vaccination against SARS CoV2 showed that the use of lower boost doses was associated with the same immunological efficacy and probably better tolerance. B cells expressing higher affinity antigen receptors being available for competition for antigen in germinal center light zones and then requiring less antigen.

Therefore we proposed that participants who received active strategies in all groups (Solo or Combi, regardless of the initial dose level received at W0,W4 and W24) be vaccinated post-W48 visit with a single 0.3 mg dose of CD40. HIVRI.Env alone or adjuvanted with Poly ICLC- Hiltonol® . This latter arm is based on preclinical CD40 vaccine data showing the good efficacy of the non-adjuvanted vaccine when delivered as a boost after initial immunizations, which will be the case for the volunteers participating in this second phase of the trial. The demonstration of a comparable effect of a booster injection with or without adjuvant is an important contribution of this trial, as the development of a non-adjuvanted protein vaccine considerably facilitates the development of such a vaccine candidate. The clinical situation (such as protection against HIV) requiring repeated booster shots to maintain a long-term memory response, the protection of which remains to be demonstrated in phase 2b/3 trials, justifies the evaluation of a non-adjuvanted booster strategy. The long-term follow-up proposed in this amendment makes it possible to evaluate long-term tolerance, maintenance of immune responses, and the effect of a distant booster injection on the maintenance of these memory responses.

Allocation of the use of the unadjuvanted vs. adjuvanted CD40. HIVRI.Env boost will be randomized. Randomisation will be stratified by the initial group (Solo or Combi with its dose level).

This second part of the trial will be single blind and consists of 3 additional visits: the late boost injection visit (WLB) and 2 follow-up visits, one 2 weeks (WLB+02) and the other 24 weeks (WLB+24) after the WLB visit.

The window for injection of the late boost is deliberately large (W48 - W76 or after, for participants who carried out the W76 visit before this amendment) as the hypothesis is that an immune memory response will be mobilized with rapid increases in post-boost immune responses, regardless of the exact timing of the late boost. This is also in line with the heterogeneous timing of late boosts in an implementation context (e.g. as is the case for current Covid-vaccine boosts, for instance).

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 65 years at the time of the screening visit (week -4)
2. Willingness and availability to be followed for the planned duration of the study in one of the dedicated investigative centers
3. Informed and signed consent
4. Agree to be registered in the French Health Ministry computerised file (for France only)
5. Being covered by the Health Insurance
6. Willingness to understake HIV testing and receive HIV test results
7. Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
8. Assessed by the clinic staff as being at "low risk" for HIV infection:

   * no history of injecting drug use in the previous ten years;
   * no STI in the last six months, untreated or incompletely treated syphilis infection in the past;
   * no high risk partner (e.g., injecting drug user, HIV positive partner) either currently or within the past six months;
   * no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known/presumed to be HIV negative;
   * no unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner.
9. Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed on the day of initial IMP administration (week 0) and before randomisation

   * Reproductive status: if heterosexually active female, consistently using an effective method of contraception with partner for sexual activity that could lead to pregnancy from at least 21 days prior to enrolment through 4 months after the last administration. Effective contraception is defined as using any of the following methods:

     * Condoms (male or female) with or without a spermicide;
     * Intrauterine device (IUD);
     * Intrauterine hormone releasing system (IUS);
     * Hormonal contraception (progesterone only);
     * Successful vasectomy in the male partner (considered successful if a participant reports that a male partner has (i) documentation of azoospermia by microscopy, or (ii) a vasectomy more than 2 years ago with no resultant pregnancy despite unprotected sexual activity postvasectomy);
     * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year without an alternative medical cause) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation.
   * Agree not to seek pregnancy including through alternative methods, such as artificial insemination or in vitro fertilization until 4 months after the last administration.
10. Participants who were born male, if heterosexually active male, using an effective method of contraception with their partner from the first day of IMP administration until 4 months after the last administration. This also applies to sperm donation.
11. Normal biological values,

    * Hemoglobin ≥ 11.0 g/dL for participants who were born female, ≥ 13.0 g/dL for participants who were born male;
    * White blood cell count = 3,300 to 12,000 cells/mm3;
    * Total lymphocyte count ≥ 800 cells/mm3;
    * Platelets = 125,000 to 550,000/mm3;
    * Chemistry panel: ALT, AST, and alkaline phosphatase < 1.25 times the institutional upper limit of normal; creatinine <1.1x institutional upper limit of normal. NB: Biological parameters outside of these values should be reviewed by the clinician who should specify the clinically significance. Results considered non-clinically significant by the clinician are accepted.
    * Negative HIV-1 and -2 blood test;
    * Negative Hepatitis B surface antigen (HBsAg);
    * Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive.
    * Normal urine test : absence of glucose, protein and hemoglobin. NB : In case of positive urinalysis dipstick results, a sample urinalysis must be performed. Results considered non-clinically significant by the clinician are accepted.

Exclusion Criteria:

1. Person participing in another research involving the human person or participing in another research involving the human person with an exclusion period still in progress at screening (week -4)
2. Intent to participate in another study of an investigational research agent during the planned duration of the study
3. Participants who are not able to understand and to follow all required study procedures for the whole period of the study in the judgment of the investigator
4. Under tutorship (only for France), guardianship, or deprived of liberty by a juridical or administrative decision
5. Planned absence that could affect participation in the study (travel abroad, relocation, impending professional mutation...)
6. Pregnant or breastfeeding
7. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

   * A process that would affect the immune response;
   * A process that would require medication that affects the immune response;
   * Any contraindication to repeated injections or blood draws;
   * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period;
   * A condition or process for which signs or symptoms could be confused with reactions to vaccine;
   * Any condition specifically listed among the exclusion criteria below.
8. Immunodeficiency
9. Asthma exclusion criteria:

   * Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).
   * Exclude a participant who:

     * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
     * Uses moderate/high dose inhaled corticosteroids, or
     * In the past year has either of the following: (i) Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids or (ii) Needed emergency care, urgent care, hospitalization, or intubation for asthma.
10. Diabetes type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes).
11. Thyroidectomy, or thyroid disease requiring medication during the last 12 months
12. Hypertension:

    * If a person has been diagnosed with hypertension, exclude for blood pressure that is not well controlled (well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic). For these participants, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrolment;
    * If a person has NOT been diagnosed with hypertension, exclude for systolic blood pressure ≥ 150 mm Hg at enrolment or diastolic blood pressure ≥ 100 mm Hg at enrolment (the measurement must be performed on a person who has been lying down for at least 5 minutes and repeated at the end of the consultation, if appropriated). Tension must be confirmed outside the clinical site to rule hypertension.
13. Contraindication to the IMPs including hypersensitivity
14. BMI ≥ 40 kg/m2 ; ≤ 18 kg/m2 ; or BMI ≥ 35 kg/m2 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
15. Bleeding disorder diagnosed by a doctor (e.g., coagulation factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
16. Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
17. Asplenia: any condition resulting in the absence of a functional spleen
18. Seizure disorder: History of seizure(s) within past three years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
19. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
20. History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including arrhythmia requiring medication, treatment, or clinical follow-up
21. History of autoimmune disease
22. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
23. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
24. Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a non-anaphylactic adverse reaction to pertussis vaccine as a child.)
25. Investigational research agents received within 30 days before first IMP administration
26. HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the investigator coordonnator will determine eligibility on a case-by-case basis.
27. Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial.
28. Live attenuated vaccines (e.g., measles, mumps, and rubella [MMR]; varicella; yellow fever) received within 30 days before first IMP administration or scheduled within 28 days after one of the 3 injections according to the protocol
29. Vaccines that are not live attenuated vaccines and were received within 21 days prior to first IMP administration (e.g., tetanus, pneumococcal, Hepatitis A or B)
30. COVID-19 vaccine received or scheduled within the last 4 weeks before and after one of the 3 injections
31. Blood products received within 120 days before first IMP administration
32. Immunoglobulin received within 60 days before first IMP administration
33. Current anti-tuberculosis (TB) prophylaxis or therapy
34. Allergy treatment with antigen injections within 30 days before first IMP administration or that are scheduled within 14 days after first IMP administration
35. Immunosuppressive medications received within last three months before first IMP administration. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrolment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Safety Part 1 - Proportion of participants without any grade 3 or 4 adverse event | Between weeks 0 and 48
  Proportion of participants without any grade 3 or 4 biological or clinical solicited local/systemic or unsolicited adverse evens, considered to be related or possibly related to IMP administration.

SECONDARY OUTCOMES:
Safety - Number of unsolicited adverse events | Between weeks 0 and 48 ; Between weeks LB and LB+24
  Overall ; by grade ; by relationship to the vaccine.
Safety - Number of solicited local and systemic adverse events | Between weeks 0 and 48 ; Between weeks LB and LB+24
  Overall ; by grade ; by relationship to the vaccine.

OTHER OUTCOMES:
Safety - Number of serious adverse events | Between weeks 0 and 48 ; Between weeks LB and LB+24
  Overall ; by grade ; by relationship to the vaccine.
Safety Part 1 - Number of Events leading to discontinuation of the vaccine regime | Between weeks 0 and 48
  Overall.
Immunological analyses : % of participants with Env-specific antibodies (Ab) | Weeks 2, 6, 26, 48 and 76; Weeks LB+2 and LB+24
  Measurement of HIV Env-specific IgG binding Ab (BAMA) against various envs and V1/V2 proteins.
Immunological analyses : Magnitude (Area under the curve) of IgG responses against Env | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of HIV Env-specific IgG binding Ab (BAMA) against various envs and V1/V2 proteins.
Immunological analyses : Breath of IgG responses against Env | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  At the highest HIV specific Ab response time point, Ab breadth will be determined using 15 additional envs panel.
Immunological analyses : % of participants with Neutralizing Ab | Weeks 2, 6, 26, 48 and 76; Weeks LB+2 and LB+24
  Measurement of Ab functionality using conventional TZM-bL neutralization assay against tier 1 and tier 2 HIV-1 isolates.
Immunological analyses : Magnitude of Neutralizing Ab (neutralizing titer, ID50) | Weeks 2, 6, 26, 48 and 76; Weeks LB+2 and LB+24
  Measurement of Ab functionality using conventional TZM-bL neutralization assay against tier 1 and tier 2 HIV-1 isolates.
Immunological analyses : Breadth of Neutralizing Ab | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of Ab functionality using conventional TZM-bL neutralization assay against tier 1 and tier 2 HIV-1 isolates.
Immunological analyses : % of lysis of reporter HIV-infected cells | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of Ab functionality using Antibody-Dependent Cell-mediated Cytotoxicity (ADCC) assay.
Immunological analyses : % of participants with B cell responses | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of Ab secretion using Elispot assay.
Immunological analyses : Magnitude of B cell responses (number of Spot Forming Units/million cells) | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of Ab secretion using Elispot assay.
Immunological analyses : % of participants with T cell responses | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of cytokine production by CD4 and CD8 T cells using Intracellular Cytokine Staining (ICS) assay.
Immunological analyses : Magnitude of the T cell response (% of cytokine-producing CD4 and CD8 T cells) | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of cytokine production by CD4 and CD8 T cells using Intracellular Cytokine Staining (ICS) assay.
Immunological analyses : % of CD4 and CD8 T cells producing 1 or more cytokine(s) | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Analysis of cell polyfunctionality using ICS.
Exploratory immunological analyses : Number of expressed genes | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Evolution of gene expression profile in the whole blood assessed by RNA Seq analysis.
Exploratory immunological analyses : Levels of cytokine secretion after specific stimulation of cells | Weeks 2, 6, 26, 48 and 76 ; Weeks LB+2 and LB+24
  Measurement of cytokine concentration in culture supernatant after specific stimulation of cells by Luminex technology.
Exploratory immunological analyses : Associations between HLA genotype and immune responses to the vaccine | Weeks 2, 6, 26 and 48
  Exploratory descriptive analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Yves LEVY, Pr, Principal Investigator — Hopital Henri Mondor
Locations (3):
- France (2):
  - Hôpital Henri Mondor, Créteil
  - CIC 1417 - Hôpital Cochin, Paris
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland